CLINICAL TRIAL: NCT01039181
Title: A Clinical Trial Phase II of Calcitriol in Combination With 5-fluorouracil, Mitomycin C and Leucovorin in an Open Label-non-randomized Study to Evaluate the Tumor Response in Patients With Advanced Intrahepatic Cholangiocarcinoma
Brief Title: Calcitriol in Advanced Intrahepatic Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Science and Technology Development Agency, Thailand (Other Government)
Collaborators: Khon Kaen University (Other)
Responsible Party: Vajarabhongsa Bhudisawasdi, Department of Surgery, Faculty of Medicine, Liver fluke and cholangiocarcinoma research center, Khon Kaen University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P-09-00171
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-12

CONDITIONS: Advanced Intrahepatic Cholangiocarcinoma
Keywords: Vitamin D; Calcitriol; cholangiocarcinoma; Clinical trial
MeSH Terms: conditions — Cholangiocarcinoma | interventions — Calcitriol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Calcitriol — 12 mcg Calcitriol will be given orally three times per week for 6 months. In this portion of the study, all patients will get the same dose of calcitriol along with the standard chemotherapy (5-fluorouracil-mitomycin C-leucovorin).
  Other Names: vitamin D

SUMMARY:
Cholangiocarcinoma (CCA), cancer of the bile duct, is the first cause of cancer death of the people in the northeast of Thailand. The incidence of CCA in this region is highest not only in the country but in the world. CCA is a slow growing but highly metastatic tumor. At present, there is no standard chemotherapy or effective treatment for CCA. Most of the patients have short survival after diagnosis. Strong evidences from in vitro, animal and clinical studies indicate that vitamin D can prevent and control growth of cancer. Our preclinical studies in CCA cell lines, animal and patient tissue culture indicate that vitamin D effectively reduce growth of CCA. Supplementation of vitamin D to chemotherapeutic drugs enhance drug toxicity and better response. At present, there are several clinical trials in USA on supplementation of vitamin D or its analogs to cancer patients. The side effect or toxicity of using vitamin D supplementation is low, some patients had stable disease and some had good response. The current study is set up a clinical trial phase II of vitamin D (calcitriol) in combination with 5-fluorouracil, Mitomycin C and Leucovorin in an open label-non-randomized study to evaluate the tumor response in patients with advanced intrahepatic cholangiocarcinoma. This study will provide an alternative/effective chemotherapy treatment for CCA patients. Better survival and improved quality of life are also expected.

DETAILED DESCRIPTION:
* OUTLINE: This is a dose-limiting toxicity study of calcitriol.
* EVALUAITON: During the initial phase, 14 patients will be accrued for this study. If the number of patient's response to calcitriol and 5-fluorouracil/mitomycin C/leucovorin is less than 1/14, the study will be stopped. However there is one patient who responses to calcitriol and 5-fluorouracil/mitomycin C/leucovorin, the new 14 patients will be accrued during the secondary phase of study.

ELIGIBILITY:
Inclusion Criteria:

1. Proven histological or cytological diagnosis of advanced intrahepatic cholangiocarcinoma (stage III, IV); Patients are ineligible for surgery.
2. Patients must have measurable or evaluable disease.
3. Age between 30-65 years
4. Performance status must be ECOG 0-1.
5. No prior use of chemotherapy or palliative radiation
6. Tumor size by CT scan must be larger than 10 mm.x10 mm.
7. Life expectancy of at least 12 weeks.
8. Adequate bone marrow, hepatic, and renal function, as evidenced by the following: WBC > 3.0 x 109/L, neutrophils > 1.5 x 109 /L; platelet count > 100 x 109/L; Hct > 30%; total bilirubin < 1 mg/dL; Liver enzymes (alkaline phosphatase, AST, ALT) < 3 times the upper limit of the normal range. Creatinine within the normal range.
9. Female patients must not be pregnant; they must be post-menopausal or practicing an accepted form of birth control. If pregnancy is a possibility, a pregnancy test will be required prior to initiation of therapy.
10. Patients must be accessible for treatment and follow-up.
11. Patient and investigator signed study-specific consent form, indicating the investigational nature of the study.

Exclusion Criteria:

1. Known hypersensitivity to Vitamin D, 5-fluorouracil, mitomycin C
2. Hypercalcemia (patients with corrected serum calcium > 10.5 mg/dL) and hyperparathyroid
3. History of renal/bladder stones
4. History of nephrectomy
5. 30 days prior to study entry, CT scan or ultrasound shows renal/bladder stones.
6. Patients with congestive heart failure or arrhythmia or unstable angina within 6 months prior study
7. Pregnancy/Lactation
8. Palliative radiation or adjuvant therapy or chemotherapy in tumor area
9. No other concurrent malignancies
10. No active infection
11. Metastasis at central nervous system
12. Metastasis at Bone
13. Renal insufficiency (creatinine > 1.5 mg/dL)
14. Patients who are in other concurrent cancer clinical trial

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-10 (Estimated); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
To assess safety and tolerability of calcitriol in combination with 5-fluorouracil/mitomycin C/leucovorin. | 3-6 months
To assess quality of life (QOL) of patients who are received calcitriol in combination with 5-fluorouracil/mitomycin C/leucovorin. | 3-6 months

SECONDARY OUTCOMES:
To assess the response of calcitriol in combination with 5-fluorouracil/mitomycin C/leucovorin in patients with advanced intrahepatic cholangiocarcinoma. | 3-6 months

CONTACTS AND LOCATIONS:
Overall Officials: Vajarabhongsa Bhudisawasdi, MD, Principal Investigator — Department of Surgery, Faculty of Medicine, Liver fluke and cholangiocarcinoma research center, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Faculty of Medicine, Khon Kaen University, Khon Kaen, Thailand

REFERENCES:
- [Derived] Sookprasert A, Pugkhem A, Khuntikeo N, Chur-in S, Chamadol N, Prawan A, Janeklang S, Vaeteewoottacharn K, Kukongviriyapan V, Pairojkul C, Bhudhisawasdi V, Wongkham S. Evaluation of efficacy, safety and tolerability of high dose-intermittent calcitriol supplementation to advanced intrahepatic cholangiocarcinoma patients--a pilot study. Asian Pac J Cancer Prev. 2012;13 Suppl:161-7. PMID 23480759